CLINICAL TRIAL: NCT00499382
Title: Quantitation of Left Ventricular Ejection Fraction as Part of F-18 FDG Whole Body PET/CT Scans For Tumor Staging
Status: Terminated | Type: Observational
Why Stopped: Slow accrual; study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0578
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Cardiac Function; Nuclear Medicine Cardiac Scan; Positron Emission Tomography; Radionuclide Ventriculography; Ventricular Ejection Fraction; PET/CT; RNV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT scan + NM cardiac scan
  Interventions: Procedure: Nuclear Medicine Cardiac Scan; Procedure: PET/CT Cardiac Scan

INTERVENTIONS:
Procedure: Nuclear Medicine Cardiac Scan — Scan lasting 30 minutes while being hooked up to a heart monitor that takes pictures every time your heart beats.
Procedure: PET/CT Cardiac Scan — Scan lasting 10-15 minutes and performed after the normally scheduled PET/CT scan.

SUMMARY:
Primary Objective:

* Evaluate the agreement between radionuclide ventriculography (RNV) and gated F-18 fluorodeoxyglucose positron emission tomography/computed tomography (FDG PET/CT) in calculating left ventricular ejection fraction (LVEF), end diastolic volume (EDV) and end systolic volume (ESV).

DETAILED DESCRIPTION:
Your doctor has ordered a PET/CT scan and a NM scan on you for routine care. By agreeing to take part in this study, you will go through both of these procedures as you normally would.

For both imaging exams, you will be lying on your back. Every effort will be made to make you as comfortable as possible. For theNM cardiac scan, you will be hooked up to a heart monitor that will take a picture every time your heart beats. Your heart will be imaged from several different views. This exam will take about 30 minutes.

The PET/CT cardiac scan will be done after completion of your normally scheduled PET/CT scan. For this scan, you will be hooked to a heart monitor that records the beats of your heart. While this monitor is attached, you will be imaged with the PET/CT scanner. The PET/CT cardiac scan will take about 10-15 minutes after your PET/CT exam is completed.

Both imaging exams will provide a number that corresponds to the percent of blood pushed out of the left ventricle of your heart during a resting state.

Taking part in this study should add between 10-15 additional minutes to your PET/CT visit. This is due to the additional cardiac imaging time.

This is an investigational study. A total of up to 50 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing both FDG PET/CT scan and RNV within two weeks interval, whether for initial staging, restaging or to evaluate response to therapy.
* Patients who would consent to an additional 10-15 minutes acquisition of the gated images after completion of their FDG PET/CT study with the additional radiation exposure.
* Patients with regular heart rate.

Exclusion Criteria:

* Blood glucose level above 200 mg/dL.
* Irregular heart rate.
* An interval of less than 1 day between the FDG PET/CT scan and RNV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with advanced cancer scheduled to have a positron emission tomography/computed tomography (PET/CT) scan and a nuclear medicine (NM) cardiac scan.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To compare the results, called an ejection fraction, of PET/CT and NM cardiac scans of heart. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Isis W. Gayed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org